CLINICAL TRIAL: NCT03553589
Title: Minimally and Non-invasive Methods for Early Detection and Progression of Endometrial Cancer
Brief Title: Biomarkers for Diagnosis and Prognosis of Endometrial Carcinoma
Acronym: BioEndoCar
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Andrea Romano (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other); Medical University of Lublin (Other)
Responsible Party: Sponsor-Investigator, Andrea Romano, PhD. Assistant Professor, Academisch Ziekenhuis Maastricht
Organization: Academisch Ziekenhuis Maastricht (Other)
Other Study IDs: NL63773
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Endometrial Cancer
Keywords: metabolomics; proteomics; early diagnosis; prognosis
MeSH Terms: conditions — Endometrial Neoplasms; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Women older than 18 years and diagnosed with endometrial cancer will be included. Blood sampling will be performed on all subjects and will be used for proteomics and metabolomics analyses.
  Interventions: Other: Blood sampling
- controls: Women older than 18 years and with a benign endometrial disturbance will be included. Blood sampling will be performed on all subjects and will be used for proteomics and metabolomics analyses.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling (10 mL) prior to standard care (e.g. surgery, medical treatment)

SUMMARY:
Endometrial cancer (EC) is the most frequent gynecological malignancy but there is currently lack of both non-invasive diagnostic tools and novel markers to stratify patients based on their risk of future recurrence. Patient care could be improved by advances in these two aspects.

In the present study, the investigators aim to identify diagnostic serum metabolite and protein biomarker signatures for early detection of cancer in asymptomatic high-risk population and prognostic biomarkers for selection of patients with poor prognosis.

DETAILED DESCRIPTION:
Rationale: Endometrial cancer (EC) is the most frequent gynaecological malignancy in the developed world. Optimal treatment of EC depends on early diagnostics and pre-operative stratification to appropriately select the extent of surgery and to plan further therapeutic approach. Currently, invasive endometrial histology is the gold standard for diagnosis, as there are no valid non-invasive methods available, and patient stratification is based on histopathology and surgical findings. There is a great need for efficient and reliable screening test for asymptomatic women with high risk of EC including Lynch syndrome patients and tamoxifen treated patients. In addition, a prognostic test is needed to stratify pre-operatively EC patients with high risk of progression in need of radical surgery together with adjuvant chemo/ratio therapy from EC patients with good prognosis. In this project the investigators are addressing this lack of non-invasive diagnostic and prognostic biomarkers of EC.

Objective: the investigators aim to identify diagnostic serum metabolite and protein biomarker signatures for early detection of cancer in asymptomatic high-risk population and (secondary objective) prognostic biomarkers for selection of patients with poor prognosis.

ELIGIBILITY:
Inclusion Criteria Cases:

* endometrioid, serous, clear cell or mucinous endometrial cancer
* dedifferentiated endometrial cancer
* high grade or low grade endometrial cancer

Inclusion Criteria Controls:

* benign uterine diseases, e.g. myoma uteri, prolapsed uterus
* prophylactic hysterectomy for Lynch syndrome

Exclusion Criteria Cases:

* atypical hyperplasia
* other types of cancer
* sarcoma uteri
* previous diagnosis of endometrial cancer

Exclusion Criteria Controls:

* any cancer
* benign ovarian diseases
* previous EC
* pregnancy at the time of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women older than 18 years and able to sign the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Creation of a diagnostic algorithm | 2020-2021
  Blood metabolome and proteome will be analysed and bioinformatics/biostatistical analysis will be used to derive diagnostic algorithms based on blood metabolites, proteins and clinical data. Algorithms in the biomarker discovery study will be developed by comparing EC and patients with benign uterine pathologies.

SECONDARY OUTCOMES:
Creation of a prognostic algorithm | 2021
  Blood metabolome and proteome will be analysed and bioinformatics/biostatistical analysis will be used to derive prognostic algorithms based on blood metabolites, proteins, clinical data at baseline and follow up information. Algorithms in the biomarker discovery study will be developed by comparing EC patients with low risk and high risk for cancer progression and recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Romano, Principal Investigator — Maastricht University Medical Centre; Tea Lanišnik Rižner, Prof. Dr., Study Chair — Faculty of Medicine, University of Ljubljana, Slovenia
Locations (5):
- Netherlands (2):
  - Maastricht University Medical Centre, Maastricht
  - Maxima Medical Centre, Veldhoven
- Lublin Medical University, Lublin, Poland
- Slovenia (2):
  - Faculty of Medicine, University of Ljubljana, Ljubljana
  - University Medical Centre, Ljubljana, Ljubljana

IPD SHARING:
Plan to Share IPD: Undecided
To be discussed within the team, put planned

REFERENCES:
- See also: Related Info — https://bioendocar.eu/